CLINICAL TRIAL: NCT00880464
Title: A Phase Ib Study of Autologous Vaccination With Lethally Irradiated, Autologous Breast Cancer Cells Engineered by Adenoviral Mediated Gene Transfer to Secrete GM-CSF Following Preoperative Chemotherapy in Women With Operable Breast Cancer
Brief Title: Autologous Vaccination With Lethally Irradiated, Autologous Breast Cancer Cells Engineered to Secrete GM-CSF in Women With Operable Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Ana C Garrido-Castro, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-216
Record Dates: First submitted 2009-04-10; First posted 2009-04-13 (Estimated); Results first posted 2021-11-09 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer
Keywords: autologous vaccination; GM-CSF; adenoviral mediated gene transfer; Stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vaccine (Experimental): Vaccinations will be administered on days 1,8,15 and every two weeks thereafter until the supply of vaccine has been exhausted or the patient is removed from study. As indicated in 5.2.5, vaccine cell dosage will be approximately 1x10 7 , 4x10 6 ,
  1x10 6 , or 1x10 5 depending on the final cell yield.
  Interventions: Biological: Autologous, Lethally Irradiated Breast Cancer Cells

INTERVENTIONS:
Biological: Autologous, Lethally Irradiated Breast Cancer Cells — Vaccination with autologous tumor cells engineered by adenoviral mediated gene transfer to secrete GM-CS

SUMMARY:
The purpose of this trial is to test the safety of a vaccine made from a patient's own breast cancer cells, and determine if this vaccine will delay or stop the growth of the cancer. The vaccine is made by genetically modifying a patient's own tumor cells to secrete granulocyte-macrophage colony-stimulating factor (GM-CSF) to activate the immune response

DETAILED DESCRIPTION:
After the patient has given their consent to participate in the trial, a series of tests will be performed to determine if the patient is eligible. These tests may take place up to 21 days before the surgery to remove a tumor sample or cancer-containing fluid, which will be used to create the vaccines. The tumor cells or fluid is then brought to a special, certified laboratory where the vaccine is made. Specially trained laboratory technicians then use a method known as adenoviral mediated gene transfer, which adds a new gene to the cancer cells. This gene causes the cells to make GM-CSF, a powerful hormone that stimulates the immune system. The cells are then given radiation so that they will not grow. Participants will start receiving vaccine on day 1, 8, 15, 29, and then every two weeks until the supply of vaccine has run out. The amount of the vaccine depends upon the total amount of cells that are obtained from the breast cancer tumor or fluid. Each time the patient is vaccinated, they will be given injections that will be placed underneath the skin. A different place will be used for each injection. If there are enough cells from the patient's tumor sample, the patient will be given an injection of non-transduced irradiated cells (the gene was not added) . These cells will help to measure how the patient's immune system is reacting to the tumor cells. This is called Delayed-Type Hypersensitivity (DTH). With vaccine #1 and #5, the patient will also receive a DTH injection. Two to three days after the vaccine and DTH injection, skin biopsies will be taken of both sites. At week 10 in the study treatment, or earlier if necessary, the patient will have a chest, abdomen, and pelvic CT scan to determine if the vaccine therapy has had an effect on their disease. A brain MRI will be performed if there were any abnormalities on the first brain MRI or if new symptoms have developed. Patients may participate in this study until one of the following happens: All vaccine created from the tumor has been given to the patient; the patient's disease worsens; the patient experiences an unacceptable and/or harmful side effect; the patient is unable to follow the study plan; or the patient's doctor feels it is no longer in the best interest of the patient to continue.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast cancer, pre-operative stages II-III per AJCC 6th edition, based on baseline evaluation by clinical examination and/or breast imaging
* Cohort 1: At least 2cm of residual disease in sum of diameters by clinical or radiographic findings following their preoperative chemotherapy
* Cohort 2: Patients who have not received preoperative chemotherapy must have at least 4cm of disease in the largest diameter by clinical or radiographic findings
* Prior therapy for Cohort 1 only: Must have completed preoperative (neoadjuvant) chemotherapy with either a standard regimen (containing an anthracycline and/or a taxane) or on a clinical trial
* HER2 positive tumors must have received at least one prior trastuzumab-based therapy, and may not receive concurrent trastuzumab therapy and vaccination
* Must initiate hormonal therapy (if indicated), including ovarian suppression, at least 4 weeks prior to initiation of vaccinations
* Must have completed definitive resection of primary tumor with adequated excision of gross disease. Surgery should have occured more than 28 days but within 12 weeks prior to enrollment
* May receive concurrent hormonal therapy, such as tamoxifen, ovarian suppression, and aromatase inhibitors
* Must have had prior banked tumor of sufficient cellular yield for vaccination
* ECOG Performance Status 0 or 1
* 18 years of age or older
* Greater than 4 weeks from immunotherapy, or systemic glucocorticoid therapy
* Adequate recovery from recent surgery and radiation therapy

Exclusion Criteria:

* Uncontrolled active infection or illness
* Other medical or psychiatric illness or social situation that would limit study compliance
* Pregnancy or nursing mothers
* Evidence of HIV infection
* Previous participation in an adenovirus-based trial
* Concurrent invasive malignancies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2011-10 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beth Overmoyer, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Anderson KS, Erick TK, Chen M, Daley H, Campbell M, Colson Y, Mihm M, Zakka LR, Hopper M, Barry W, Winer EP, Dranoff G, Overmoyer B. The feasibility of using an autologous GM-CSF-secreting breast cancer vaccine to induce immunity in patients with stage II-III and metastatic breast cancers. Breast Cancer Res Treat. 2022 Jul;194(1):65-78. doi: 10.1007/s10549-022-06562-y. Epub 2022 Apr 28. PMID 35482127

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2006 through May 2008
Groups:
- Stage II-III Breast Cancer Cohort: Biological/Vaccine: Autologous, Lethally Irradiated Breast Cancer Cells Vaccine will be administered on days 1, 8, 15, 29 and then every 2 weeks until the supply of vaccine runs out
  Autologous, Lethally Irradiated Breast Cancer Cells: Vaccination with autologous tumor cells engineered by adenoviral mediated gene transfer to secrete GM-CS
Period: Overall Study
Arm/Group | Stage II-III Breast Cancer Cohort
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Metastatic Breast Cancer Cohort: Biological/Vaccine: Autologous, Lethally Irradiated Breast Cancer Cells Vaccine will be administered on days 1, 8, 15, 29 and then every 2 weeks until the supply of vaccine runs out
  Autologous, Lethally Irradiated Breast Cancer Cells: Vaccination with autologous tumor cells engineered by adenoviral mediated gene transfer to secrete GM-CS
Arm/Group | Metastatic Breast Cancer Cohort
Number analyzed (Participants) | 7
Age, Continuous [Mean (Full Range); unit: years] | 51.5 [32 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Clinical Stage [Count of Participants; unit: Participants] — T1: tumor is 2 cm or less T2 tumor is between 2 and 5 cm T3: tumor is greater than 5 cm T4: tumor has spread into the the chest wall and/or skin
  N0: no tumor in lymph nodes N1: tumor(s) in axillary lymph nodes N2: tumor(s) in axillary lymph nodes fixed of matted or only in clinically apparent mammary nodes without clinically evident axillary lymph nodes.
  N3: tumor(s) in infraclavicular lymph nodes or clinically apparent internal mammary lymph nodes or supraclavicular lymph nodes
  M0: cancer hasn't spread to other parts of the body M1: cancer has spread to other parts of the body
  Participants
    T3, N1 | 3
    T4, N0, M1 | 1
    T4, N1 | 2
    T4, N2 | 1
Hormone Receptor Status [Count of Participants; unit: Participants]
  Positive | 5
  Negative | 2
Human Epidermal Growth Factor Receptor 2 Status [Count of Participants; unit: Participants]
  Positive | 1
  Negative | 6
Triple Negative [Count of Participants; unit: Participants]
  Positive | 2
  Negative | 5
Type of Surgery [Count of Participants; unit: Participants]
  Mastectomy | 6
  Lumpectomy | 1
Pathologic Response to Neoadjuvant Therapy [Count of Participants; unit: Participants]
  Partial Response | 6
  Not Available | 1

OUTCOME MEASURES:

1. Primary Outcome: Minimum Number of Vaccine Doses Created Using Participant Tumor Sample
Description: Tumor samples were obtained via malignant effusion or a surgically accessible tumor nodule of 2 cm in greatest diameter. Tumor cells were processed to single cell suspension and transduced with adenoviral vector encoding human Granulocyte-macrophage colony-stimulating factor (GM-CSF). Then, the cells washed extensively and irradiated with 10,000 cGy. Over the next 14 days, sterility cultures were tested for endotoxin and mycoplasma contamination. Individual vaccine cell dose and number varied depending on the final cell yield from vaccine production. For stage II-III patients, the minimal dose was 1 x 10^5 cells and the maximal dose was 4 x 10^6 cells. For metastatic patients, the minimal dose was 1 x 10^5 cells and the maximal dose was 1 x 10^7 cells.
Time Frame: 40 Months
Population: Vaccinations prepared for "enrolled for vaccine administration" population.
Measure: Number; unit: doses
Groups:
- Vaccine: Biological/Vaccine: Autologous, Lethally Irradiated Breast Cancer Cells Vaccine will be administered on days 1, 8, 15, 29 and then every 2 weeks until the supply of vaccine runs out
  Autologous, Lethally Irradiated Breast Cancer Cells: Vaccination with autologous tumor cells engineered by adenoviral mediated gene transfer to secrete GM-CS
Arm/Group | Vaccine
Number analyzed (Participants) | 7
doses | 6

2. Primary Outcome: Number of Participants With Grade 3 or Higher Adverse Events
Description: Number of participants with grade 3 or higher adverse events as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Up to 58 Months
Population: Analysis population for adverse events is "Treated" population.
Measure: Count of Participants; unit: Participants
Arm/Group | Vaccine
Number analyzed (Participants) | 7
Participants
  Grade 3 | 1
  Grade 4 | 0
  Grade 5 | 0

3. Secondary Outcome: Median Follow-up Time by Survival Status
Description: Participants followed for survival status. Participants who were alive were noted as such as late as December 2020.
Time Frame: Up to 14 Years
Population: Clinical outcomes assessed for the "treated" population.
Measure: Median (Full Range); unit: years
Arm/Group | Vaccine
Number analyzed (Participants) | 7
years
  Alive: number analyzed (Participants) | 2
  Alive | 9.88 [9.76 to 9.99]
  Dead: number analyzed (Participants) | 5
  Dead | 6.24 [1.16 to 8.49]

ADVERSE EVENTS:
Time Frame: Up to 14 Years
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Vaccine
All-Cause Mortality (participants affected / at risk) | 5/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=7)
Fatigue (General disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (N=7)
Allergic Reaction (Immune system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Fat atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Fatigue (General disorders) | 7 (17)
Fever (General disorders) | 2 (2)
Headache (Nervous system disorders) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)
Hot Flashes (Vascular disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (7)
Memory Impairment (Nervous system disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (3)
Pain (General disorders) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes